CLINICAL TRIAL: NCT04273399
Title: Feasibility of High-impact Exercise to Improve Musculoskeletal Outcomes in Adults With Crohn's Disease
Brief Title: High-impact Exercise in Adults With Crohn's Disease
Acronym: IMPACT CD
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: NHS Greater Glasgow and Clyde (Other)
Collaborators: University of Glasgow (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GN19GA462
Record Dates: First submitted 2020-01-08; First posted 2020-02-18 (Actual); Last update posted 2020-02-18 (Actual); Status verified 2020-02

CONDITIONS: Crohn Disease
Keywords: Crohn's Disease; Exercise; Feasibility
MeSH Terms: conditions — Crohn Disease; Motor Activity

STUDY DESIGN:
Intervention Model Description: Case control model
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Crohn's Disease (Experimental): Twelve week jumping based exercise intervention
  Interventions: Other: High-impact exercise intervention; Other: Acute response to high-impact exercise
- Controls (Active Comparator): Age and sex matched controls will undertake the same twelve week intervention for active comparison between groups
  Interventions: Other: High-impact exercise intervention; Other: Acute response to high-impact exercise

INTERVENTIONS:
Other: High-impact exercise intervention — * Twelve-week high-impact exercise intervention
  * Majority home based sessions, some supervised sessions
  * Three exercise sessions per week
  * Between 50 - 100 jumps per session
  * Progressive jumping exercises to increase mechanical loading
Other: Acute response to high-impact exercise — * First session of twelve-week high-impact exercise session used to assess the acute physiological response to one session of high-impact exercise in both Crohn's disease and healthy controls
  * One supervised session of high-impact exercise
  * Bloods to assess acute inflammatory and bone turnover response post-exercise

SUMMARY:
Crohn's disease increases the risk of poor musculoskeletal health, as the inflammatory disease process directly inhibits regulatory pathways involved in bone and muscle formation and maintenance. The negative effects of disease on muscle-bone health are compounded by poor nutritional status, vitamin d deficiency, prolonged exposure to glucocorticoid therapy, and reduced physical activity. Modern, steroid sparing therapies are successful at inducing clinical remission in terms of inflammation, however they have limited effect in remedying observed muscle-bone deficits. Subsequently, patients with Crohn's disease are at increased lifelong risk of pathological fractures and osteoporosis. Novel adjunctive therapies are therefore required to complement pharmacological treatments and target muscle-bone deficits, which are responsible for significant disease burden in Crohn's.

High-impact exercise may be a useful additional therapy for patients with Crohn's disease, as the mechanical strains produced during this type of exercise, through large magnitude muscular contractions and ground reaction forces, can promote bone formation and gains in muscle mass. There have been no previous studies assessing the effects of high impact exercise in Crohn's disease, so it is unknown if this type of exercise is safe and feasible in this population. The aim of this study is to assess the feasibility of high-impact exercise for improving markers of bone and muscle health in adults with Crohn's disease, and compare the effects of exercise with a group of healthy age and sex matched controls.

ELIGIBILITY:
Inclusion Criteria:

* Crohn's disease diagnosed at least six months ago
* Stable medication for at least four weeks
* Disease in remission, or mildly/moderately active according to Harvey Bradshaw Index score
* Currently undertaking <2 hours of structured exercise per week
* Able to mobilise and exercise independently
* Able to provide written informed consent

Exclusion Criteria:

* Surgery <12 weeks or planned surgery during intervention period
* Comorbidity known to affect muscle / bone
* Contraindication to high-impact exercise
* Pregnancy or planned pregnancy during intervention period
* BMI >40 kg/m2 (or body mass >120kg)

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2020-03 (Estimated); Primary Completion 2021-10 (Estimated); Study Completion 2021-10 (Estimated)

PRIMARY OUTCOMES:
Feasibility of participation in high-impact exercise: proportion of exercise sessions completed, and proportion of repetitions completed across intervention | Through intervention period (4 weeks).
  Adherence to exercise intervention - measured as proportion of exercise sessions completed, and proportion of repetitions completed across intervention.

SECONDARY OUTCOMES:
Change in Tibia Bone Density & Geometry | Assessed at baseline (pre-intervention) and follow up (<14 days post-intervention)
  Peripheral quantitative computed tomography (pQCT)
Change in Whole Body Bone Density & Composition | Assessed at baseline (pre-intervention) and follow up (<14 days post-intervention)
  Dual energy x-ray absorptiometry scan
Change in Inflammatory Cytokines | Intervention effects: Bloods measured at baseline (pre-intervention), midpoint of intervention (Week 7) and <7 days post-intervention to assess changes. Acute effects of exercise: measured pre-exercise, then 0, 15, 30 and 60 minutes post-exercise
  Pro-inflammatory cytokines in blood (Interleukin [IL-] 1Beta, IL-6, IL-17, Tumour necrosis factor alpha) [all in pg/ml]
Change in Bone Formation Marker | Intervention effects: Bloods measured at baseline (pre-intervention), midpoint of intervention (Week 7) and <7 days post-intervention to assess changes. Acute effects of exercise: measured pre-exercise, then 0, 15, 30 and 60 minutes post-exercise
  Bone specific alkaline phosphatase [ug/ml]
Change in Bone Resorption Marker | Intervention effects: Bloods measured at baseline (pre-intervention), midpoint of intervention (Week 7) and <7 days post-intervention to assess changes. Acute effects of exercise: measured pre-exercise, then 0, 15, 30 and 60 minutes post-exercise
  C-telopeptide of type I collagen and Sclerostin [both ng/ml]
Change in Disease Specific Health related quality of life | Assessed at baseline (pre-intervention), mid-point of intervention (Week 7) and follow up (<7 days post-intervention). Scale 32 - 224; higher score means better quality of life.
  Inflammatory Bowel Disease Questionnaire (CD Group Only)
Change in Health related quality of life | Assessed at baseline (pre-intervention), mid-point of intervention (Week 7) and follow up (<7 days post-intervention). Scale 0 to 100, higher score equals better quality of life.
  PedsQL Generic Core Scale (CD & Control group)
Change in disease related Fatigue | Assessed at baseline (pre-intervention), mid-point of intervention (Week 7) and follow up (<7 days post-intervention). Scale 0 - 120, lower score equals less problems with fatigue.
  Inflammatory Bowel Disease Fatigue questionnaire (CD Group)
Change in Fatigue | Assessed at baseline (pre-intervention), mid-point of intervention (Week 7) and follow up (<7 days post-intervention). Scale 0 - 100, higher score equals less problems with fatigue.
  Multidimensional Fatigue Scale (CD & Control group)
Change in Lower limb muscle function | Assessed at baseline (pre-intervention), mid-point of intervention (Week 7) and follow up (<7 days post-intervention)
  Jumping Mechanography
Habitual physical activity | Seven days post-baseline visit.
  Wrist-worn accelerometry
Self-efficacy for exercise: questionnaire | Pre-intervention. Self-efficacy for exercise scale: Nine-item scale, score 0-10 per item. Min value 0, Max Value 90. Higher score equals better self-efficacy.
  Self-efficacy for exercise questionnaire
Change in Disease activity | Assessed at baseline (pre-intervention), mid-point of intervention (Week 7) and follow up (<7 days post-intervention). Scale 0 to >450. Score 0-150 = remission, 151-220 = mild disease, 220-450 = moderate disease, >450 = severe disease.
  Crohn's disease activity index (CD only)
Change in Dietary Intake | Assessed at baseline (pre-intervention), mid-point of intervention (Week 7) and follow up (<7 days post-intervention)
  Three-day estimated weight food diary
Change in Body composition | Assessed at baseline (pre-intervention), mid-point of intervention (Week 7) and follow up (post-intervention)
  Bio-electrical impedance (Body mass, Fat Mass, Fat Free Mass [all in kg])
Changes in Inflammatory marker in stool sample | Assessed at baseline (pre-intervention), mid-point of intervention (Week 7) and follow up (post-intervention)
  Faecal Calprotectin (ug/g)

CONTACTS AND LOCATIONS:
Overall Officials: Jarod Wong, Principal Investigator — NHS Greater Glasgow & Clyde
Locations (1):
- Queen Elizabeth University Hospital, NHS Greater Glasgow & Clyde, Glasgow, United Kingdom

IPD SHARING:
Plan to Share IPD: No